CLINICAL TRIAL: NCT01994343
Title: Musculoskeletal Disturbances in Women With Chronic Pelvic Pain
Brief Title: Pain in Women With Chronic Pelvic Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, Marie Carmen Valenza, assistant professor, Universidad de Granada
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DF0044UG
Record Dates: First submitted 2013-11-19; First posted 2013-11-25 (Estimated); Last update posted 2018-07-24 (Actual); Status verified 2018-07

CONDITIONS: Chronic Pain
Keywords: Chronic pelvic pain, women, pain, posture.
MeSH Terms: conditions — Chronic Pain; Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Experimental group (Experimental): Adult women aged over 18 years old with pain during more than six months are included in the study. These patients will receive a global posture reeducation.
  Interventions: Other: Global posture reeducation
- Control group (No Intervention): Adult women aged over 18 years old without chronic pain. will receive no intervention.

INTERVENTIONS:
Other: Global posture reeducation — An assessment of the women is performed using global posture reeducation.
  Other Names: Evaluation
  Arms: Experimental group

SUMMARY:
Chronic pelvis pain is very common between adult women. Significant progress is made in clarifying the multifactorial model of chronic pain pathogenesis, but a more complete assessment is important in order to improve the therapeutic approach. The purpose of this study is stablish a clinical and symptomatological profile of women with chronic pelvic pain.

DETAILED DESCRIPTION:
Chronic pelvic pain is defined as non-menstrual or noncyclic pelvic pain with duration of at least 6 months. This pain interfere with habitual activities and requires clinical or surgical treatment. It is a complex interaction between the gastrointestinal, urinary, gynecologic, musculoskeletal, neurologic and endocrine systems influenced by psychological factors. Its prevalence range between 3 and 8% among women aged 15-73 years, ranging from 14 to 24% among women of reproductive age. It is very important a multidimensional approach in order to stablish a more specific profile.

ELIGIBILITY:
Inclusion Criteria:

* Women.
* Clinical diagnosis of chronic pelvic pain.
* More than eighteen years.
* Non-menstrual or noncyclic pelvic pain.
* Duration of pain of at least 6 months.

Exclusion Criteria:

* Duration of pain less than 6 months.
* Women who were pregnant in the last 12 months

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2013-11; Primary Completion 2016-12 (Actual); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
Change in postural control | Change from baseline postural control at 8 weeks
  Postural control will be assessed using the Mini-BESTest, a 14-item test that focuses on dynamic balance, specifically anticipatory transitions (six items), reactive postural control (six items), sensory orientation (six items), and dynamic gait (10 items). Each item is scored from 0 to 2; a score of 0 indicates that a person is unable to perform the task, whereas a score of 2 is normal. The best score is the maximum amount of points, being 28.

SECONDARY OUTCOMES:
Nervous assessment | baseline
  The nervous assessment is measured with neurodynamic tests. This is used to test upper and lower extremities. It moves most of the nerves between the neck and legs, including the spinal nerves and lower limbs nerves.
  The patient is placed in supine position. It is measured with a goniometer.
Spinal assessment | baseline
  The spinal assessment is going to be performed using the Spinal Mouse. Spinal Mouse is a device that, combined with a computer program, assesses the curvatures of the vertebral column without applying harmful radiation. Spinal Mouse checks: spine alignment, measuring segmental and global angles in the sagittal and frontal planes; posture and spinal mobility; spine functions and performance.
Balance under dual task conditions | Baseline, 8 weeks
  Women were asked to complete three trials of the TUG under three conditions: performance of the TUG alone, performance of the TUG with the addition of a cognitive task (TUG cognitive), and performance of the TUG with the addition of an upper-extremity motor task (TUG manual). Women were given verbal instructions to stand up from a chair, walk 3 m as quickly and as safely as possible, cross a line marked on the floor, turn around, walk back, and sit down. In the TUG cognitive, women were asked to complete the test while counting backward by threes from a randomly selected number between 20 and 100. In the TUG manual, women were asked to complete the test while carrying a full cup of water.
Trigger points evaluation | baseline
  Trigger points are discrete, focal, hyperirritable spots located in a taut band of skeletal muscle. A pressure at a trigger point is performed in order to evoke pain at the point as well as referred pain in myofascial or visceral structures. The trigger points located in the gluteal and adductors muscles are going to be assessed.
Self perceived health status | Baseline, 8 weeks.
  Health status was assessed by the Euroqol-5dimensions (EQ-5D). It is divided into 2 sections. The first section contains 5 questions about mobility, self-care, usual activities, pain/discomfort and anxiety/depression. For each question, problems within the domain are evaluated on a 3-level basis. Responders can choose between "no problems", "some problems" or "extreme problems". The second part is a visual analogue scale (VAS) score, which records the responder's self-evaluated health status, where 0 is worst imaginable health and 100 is best imaginable health.

CONTACTS AND LOCATIONS:
Overall Officials: Marie Carmen Valenza, PhD, Principal Investigator — Universidad de Granada
Locations (1):
- Department of Physical Therapy, Granada, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Rodriguez-Torres J, Lopez-Lopez L, Cabrera-Martos I, Prados-Roman E, Granados-Santiago M, Valenza MC. Effects of an Individualized Comprehensive Rehabilitation Program on Impaired Postural Control in Women With Chronic Pelvic Pain: A Randomized Controlled Trial. Arch Phys Med Rehabil. 2020 Aug;101(8):1304-1312. doi: 10.1016/j.apmr.2020.02.019. Epub 2020 Apr 20. PMID 32325162
- [Derived] Fuentes-Marquez P, Valenza MC, Cabrera-Martos I, Rios-Sanchez A, Ocon-Hernandez O. Trigger Points, Pressure Pain Hyperalgesia, and Mechanosensitivity of Neural Tissue in Women with Chronic Pelvic Pain. Pain Med. 2019 Jan 1;20(1):5-13. doi: 10.1093/pm/pnx206. PMID 29025041